CLINICAL TRIAL: NCT01859130
Title: Persona Outcomes Led Assessment Research in Total Knee Arthroplasty
Brief Title: Zimmer POLAR - Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSU2012-10K
Record Dates: First submitted 2013-05-16; First posted 2013-05-21 (Estimated); Results first posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis; RheumatoId Arthritis; Traumatic Arthritis; Polyarthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Persona TKA (Other): Primary total knee arthroplasty subjects that receive the Zimmer Persona Total Knee System
  Interventions: Device: Zimmer Persona Total Knee System

INTERVENTIONS:
Device: Zimmer Persona Total Knee System
  Other Names: Primary Knee Replacement,; Total Knee Arthroplasty,; Total Knee Replacement

SUMMARY:
The primary objective of this study is to obtain implant survivorship and clinical outcomes data for commercially available Persona fixed bearing knee implants used in total knee arthroplasty. The assessment will include implant survivorship and clinical performance measured by pain and function, quality of life data, radiographic parameters and survivorship.

DETAILED DESCRIPTION:
The study design is a prospective, multicenter, study of the commercially available Persona fixed bearing knee implants. The study will require each site to obtain Institutional Review Board (IRB) approval prior to study enrollment. All potential study subjects will be required to participate in the Informed Consent Process.

All study subjects will undergo preoperative clinical evaluations prior to their total knee arthroplasty. The post-operative clinical and radiographic evaluations will be conducted at 6 weeks, 6 months, 1 year, 2, 3, 4, and 5 years.

All info specified in the Brief Summary will be captured via the Knee Society Score, EQ-5D, Forgotten Joint Score, KSS Patient Expectations, Physical Exam, and Physician's Assessment of Radiographic Outcomes form.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18-75 years of age, inclusive;
* Patient qualifies for primary total knee arthroplasty based on physical exam and medical history, including diagnosis of severe knee pain and disability due to at least one of the following:

  * rheumatoid arthritis, osteoarthritis, traumatic arthritis, polyarthritis;
  * collagen disorders and/or avascular necrosis of the femoral condyle;
  * post-traumatic loss of joint configuration, particularly when there is patellofemoral erosion, dysfunction or prior patellectomy;
  * moderate valgus, varus, or flexion deformities;
  * the salvage of previously failed surgical attempts that did not include partial or total knee arthroplasty of the ipsilateral knee;
* Patient has participated in a study-related Informed Consent process;
* Patient is willing and able to complete scheduled study procedures and follow-up evaluations;
* Independent of study participation, patient is a candidate for commercially available Persona fixed bearing knee components implanted in accordance with product labeling.

Exclusion Criteria:

* Patient is currently participating in any other surgical intervention studies or pain management studies;
* Previous history of infection in the affected joint and/or other local/systemic infection that may affect the prosthetic joint;
* Insufficient bone stock on femoral or tibial surfaces;
* Skeletal immaturity;
* Neuropathic arthropathy;
* Osteoporosis or any loss of musculature or neuromuscular disease that compromises the affected limb;
* Stable, painless arthrodesis in a satisfactory functional position;
* Severe instability secondary to the absence of collateral ligament integrity;
* Rheumatoid arthritis accompanied by an ulcer of the skin or a history of recurrent breakdown of the skin;
* Patient has a known or suspected sensitivity or allergy to one or more of the implant materials;
* Patient is pregnant or considered a member of a protected population (e.g., prisoner, mentally incompetent, etc.);
* Patient has previously received partial or total knee arthroplasty for the ipsilateral knee.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2013-10-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kacy Arnold, RN MBA, Study Director — Zimmer Biomet
Locations (4):
- United States (4):
  - Midwest Orthopaedics at Rush, Naperville, Illinois
  - The Rothman Institute, Egg Harbor, New Jersey
  - Duke University, Durham, North Carolina
  - The Rothman Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Persona TKA: Primary total knee arthroplasty subjects that receive the Zimmer Persona Total Knee System
  Zimmer Persona Total Knee System
Period: Overall Study
Arm/Group | Persona TKA
Started | 299
Completed | 192
Not Completed | 107
Not completed — Death | 4
Not completed — Lost to Follow-up | 16
Not completed — Sponsor terminated: 47 Not specified: 3 | 53
Not completed — Physician Decision | 6
Not completed — Withdrawal by Subject | 17
Not completed — Adverse Event | 11

BASELINE CHARACTERISTICS:
Population: Patient demographics were captured for 326 subjects, however 27 subjects were study completed prior to surgery and prior to pre-op Patient Report Outcome Measure Completion. Therefore, 299 are included in this submission.
Arm/Group | Persona TKA
Number analyzed (Participants) | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 153
  >=65 years | 146
Age, Continuous [Mean (Full Range); unit: years] | 62.88 [44 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157
  Male | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 296
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 299
EQ5D-5L [Mean (Full Range); unit: units on a scale] — Each EQ-5D comprises a short descriptive questionnaire and a visual analogue scale (EQ VAS). The questionnaire provides a simple descriptive profile of a respondent's health state. The EQ VAS provides an alternative way to elicit an individual's rating of the individual's own overall current health. The overall range is -0.1 to 1.0. A higher score indicates a better overall health rating reported by the patient, and a lower score indicates a poor overall health rating. It is possible to score a negative value. Although unlikely, a negative value is observed to be a state worse than death. Population: Patient demographics were captured for 326 subjects, however 27 subjects were study completed prior to surgery and prior to pre-op Patient Report Outcome Measure Completion. All other analyses will include 299 subjects (beginning with PROMs).
  units on a scale | 0.5 [-0.1 to 1.0]
Knee Society Score - Objective Knee [Mean (Full Range); unit: units on a scale] — This form includes alignment, instability, joint range of motion, and symptoms. The overall scoring range is -8 to 106. A higher score indicates good alignment, range of motion, and minimal symptoms of pain. A lower score indicates poor knee alignment, potential issues in range of motion, and the very likely experience of symptoms of pain. Population: Patient demographics were captured for 326 subjects, however 27 subjects were study completed prior to surgery and prior to pre-op Patient Report Outcome Measure Completion. All other analyses will include 299 subjects (beginning with PROMs).
  units on a scale | 47.3 [-8.0 to 96.0]
KSS Patient Expectations [Mean (Full Range); unit: units on a scale] — This is a 3 question form to evaluate a patient's expectations of their knee replacement prior to receiving it. This score serves as the baseline to measure how expectations were met postoperatively. The overall score possibility ranges from 3 to 15. A score of 3 would indicate that the patient has very low expectations for surgery, and a score of 15 would indicate that the patient has very high expectations for surgery in terms of relief of pain, performing normal activities, and performing recreational activities. Population: Patient demographics were captured for 326 subjects, however 27 subjects were study completed prior to surgery and prior to pre-op Patient Report Outcome Measure Completion. All other analyses will include 299 subjects (beginning with PROMs).
  units on a scale | 14.4 [9.0 to 15.0]

OUTCOME MEASURES:

1. Primary Outcome: Knee Society Scores
Description: This form includes alignment, instability, joint range of motion, and symptoms. The overall range of scores available is -8 to 106. A higher score indicates good alignment, range of motion, and minimal symptoms of pain. A lower score indicates poor knee alignment, potential issues in range of motion, and the likely experience of symptoms of pain.
Time Frame: 5 years post op
Population: Only 161 subjects completed the KSS form at the final 5yr follow-up. All other subjects were study completed, or lost to follow-up.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Persona TKA
Number analyzed (Participants) | 161
units on a scale | 92.9 [57.0 to 102.0]

2. Secondary Outcome: EQ-5D
Description: The EQ-5D family of instruments has been developed to evaluate health across a wide range of disease areas. Each EQ-5D instrument comprises a short descriptive system questionnaire and a visual analogue scale (EQ VAS). The questionnaire provides a simple descriptive profile of a respondent's health state. The EQ VAS provides an alternative way to elicit an individual's rating of the individual's own overall current health. The overall range is -0.1 to 1.0. A higher score indicates a better overall health rating reported by the patient, and a lower score indicates a poor overall health rating. It is possible to score a negative value. Although unlikely, a negative value is observed to be a state worse than death.
Time Frame: 5 years post op
Population: Only 175 subjects completed the EQ-5D form at the final 5yr follow-up. All other subjects were study completed, or lost to follow-up.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Persona TKA
Number analyzed (Participants) | 175
units on a scale | 0.9 [-0.0 to 1.0]

3. Secondary Outcome: Forgotten Joint Score (FJS)
Description: The Forgotten Joint Score-12 (FJS-12) is a validated patient-reported outcome measure (PROM) tool designed to assess artificial prosthesis awareness during daily activities following total knee arthroplasty (TKA). Scores range from 0-100. A score of 100 would indicate a high degree of "forgetting" the artificial joint (a low degree of awareness). A score of 0 would indicates a very low degree of "forgetting" the artificial joint (typically aware of the replacement).
Time Frame: 5 years post-op
Population: Only 176 subjects completed the FJS form at the final 5yr follow-up. All other subjects were study completed, or lost to follow-up.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Persona TKA
Number analyzed (Participants) | 176
units on a scale | 74.9 [0.0 to 100.0]

ADVERSE EVENTS:
Time Frame: Postoperatively through study completion (5yr follow-up).
Arm/Group | Persona TKA
All-Cause Mortality (participants affected / at risk) | 4/299
Serious Adverse Events (participants affected / at risk) | 72/299
Other Adverse Events (participants affected / at risk) | 227/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Persona TKA (N=299)
Cardiovascular (Cardiac disorders) | 11 (12) — Chest pain Chest pressure Congestive Heart Failure Atrial Fibrillation
Generic Cardiovascular Reports (Cardiac disorders) | 3 (3) — Cerebral Ischemic Stroke Blockage in Artery DX of SVT
Dermatological Disorders (Skin and subcutaneous tissue disorders) | 3 (3) — Hives and rashes Cellulitis left shin
Adrenal insufficiency (Metabolism and nutrition disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 5 (5) — Appendicitis Gall Bladder Bleeding ulcers Colon resection
Genitourinary / Renal (Renal and urinary disorders) | 5 (5)
Hematological (Blood and lymphatic system disorders) | 1 (1)
Infection (non-knee) (Infections and infestations) | 3 (3)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 26 (26)
Neurological (Nervous system disorders) | 7 (8)
Oncological (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Pulmonary / Respiratory (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Wound Drainage / Device Loosening (Surgical and medical procedures) | 2 (2)
Other General Adverse Events (General disorders) | 10 (12)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Persona TKA (N=299)
Gastrointestinal (Gastrointestinal disorders) | 41 (47)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 145 (246)
Other General Adverse Events (General disorders) | 118 (180)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT01859130/Prot_SAP_000.pdf